CLINICAL TRIAL: NCT03473418
Title: Ketoconazole In Situ Gel Versus Terconazole Cream for Treatment of Vaginal Candidiasis
Brief Title: Ketoconazole Gel Versus Terconazole Cream for Vaginal Candidiasis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariana Noss Abdo, Egypt Assiut ( Elghnium city), Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KTVC
Record Dates: First submitted 2018-03-04; First posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Vaginal Candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Ketoconazole; terconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketoconazole gel (Experimental): use of Ketoconazole in situ gel for treatment of vaginal candidiasis
  Interventions: Drug: Ketoconazole
- terconazole cream (Active Comparator): use of terconazole 0.8 cream for treatment of vaginal candidiasis
  Interventions: Drug: Terconazole

INTERVENTIONS:
Drug: Ketoconazole — Ketoconazole as a topical vaginal gel
  Arms: Ketoconazole gel
Drug: Terconazole — Terconazole 80 mg as a topical vaginal cream
  Arms: terconazole cream

SUMMARY:
Vaginal Candidiasis is an infection caused by a yeast normally lives inside the body . Sometimes Candida can multiply and cause an infection if the environment inside the vagina changes in a way that encourages its growth. Candidiasis in the vagina is commonly called a "vaginal yeast infection." Risk factor use of intra uterine devices , pregnancy ,use hormonal contraceptives ,have diabetes , immune compromised taken antibiotics Diagnosis cause itching or soreness Pain during sexual intercourse Pain or discomfort when urinating and abnormal vaginal discharge Although most vaginal candidiasis is mild, some women can develop severe infections involving redness, swelling, and cracks in the wall of the vagina

DETAILED DESCRIPTION:
terconazole- Terconazole, an azole antifungal agent, inhibits fungal cytochrome P-450-mediated 14 alpha-lanosterol demethylase enzyme. This enzyme functions to convert lanosterol to ergosterol. The accumulation of 14 alpha-methyl sterols correlates with the subsequent loss of ergosterol in the fungal cell wall and may be responsible for the antifungal activity of Terconazole. Mammalian cell demethylation is less sensitive to Terconazole inhibition Terconazole exhibits antifungal activity in vitro against Candida albicans and other Candida species. The MIC (maximum insufflation capacity values of Terconazole against most Lactobacillus spp. typically found in the human vagina were ≥128 mcg/mL; therefore these beneficial bacteria are not affected by drug treatment.

Terconazole Vaginal cream, 80 mg are indicated for the local treatment of vulvovaginal candidiasis (moniliasis). As this product is effective only for vulvovaginitis caused by the genus Ketoconazole is a broad- spectrum antimycotic agent that can be used orally or topically in the treatment vulvovaginal candidiasis and other fungal infections Candida is the second most common cause of vaginal infections. Candida albicans is responsible for 80 to 92% of episodes of vulvovaginal candidiasis . The rest are due to non-albicans Candida species, the most common of which are C. glabrata and C. tropicalis. Sporadic attacks of vulvovaginal candidiasis usually occur without an identifiable precipitating factor. The risk of vulvovaginal candidiasis may be higher in women with uncontrolled diabetes, who use oral contraceptives containing high levels of estrogen or taking antibiotics.

In situ gelling systems refer to polymer solutions which can be administered as liquid, and undergo a phase transition to semisolid gel upon exposure to physiological environments. Stimuli- sensitive hydrogels are those hydrogels, which undergo reversible volume phase - transition or sol - gel phase transition in response to external physical stimuli such as (temperature) or chemical stimuli as (ions).The most commonly used thermoreversible gels are those prepared from the pluronic block copolymers . The principle advantage of in situ forming gels is the possibility of administering accurate and reproducible quantities, in contrast to already gelled formulation . Several in situ gel forming systems have been developed to prolong the residence time of a drug and improve the bioavailability and control the drug release by changing the gel structure in response to environmental stimuli . These systems provide simplicity and safety in in vivo situations . They are handled in the liquid state before their delivery, which is likely to facilitate their use and to increase the surface of contact with the mucous membrane. The flow properties of semi-solid vaginal dosage forms might be of use to predict the spreading and coating of the formulations over the vaginal epithelia . When the preparation is given as liquid, this will give better spreading and coating of vaginal surfaces than the gelled preparations, which have not the ability to cover all the surfaces and cannot reach to epithelial folds of the vagina. So, this study aimed to formulate ketoconazole in a new vaginal mucoadhesive form "In situ gel" and it is designed to achieve the following objectives:

* Formulation and evaluation of in situ-forming vaginal gels of ketoconazole.
* Clinical assessment of the prepared vaginal ketoconazole in situ gels on women suffering from vaginal candidiasis.

Materials and Methods:

Preparation of ketoconazole vaginal in situ gel Different concentrations of pluronic F-127 will be used in the preparation of the in situ forming gels. Medicated in situ forming gels will be prepared on a weight basis using The Modified Cold Method .Vaginal preparations will be prepared in citro-phosphate buffer pH (power of hydrogen) 4.5.

Characterization of ketoconazole vaginal in situ gel

* Gelation temperature (Tgel) measurement Ten milliliters of cold pluronic solution and a magnetic bar will be put into a beaker (25 ml) that will be placed in a low temperature water bath at room temperature. A thermometer will be immersed in the sample solution. The solution will be heated at constant rate with continuous stirring at a rate of 200 rpm. The temperature at which the magnetic bar stopped to move due to gelation will be reported as the gelation temperature (Tgel) (11).
* Rheological studies The viscosity of each formula will be determined using a Brookfield DV (diluted volume )-III Ultra viscometer (RV model). The spindles used will be 60 for liquids and 95 for gels. Measurements will be carried out at spindle speed of 15 rpm. Viscosity will be measured at different temperatures 4ºC (celsius degree ), 25ºC, and 37ºC.
* In vitro release of Ketoconazole from in situ gelling formulations In vitro release from in situ gelling formulae will be studied using a standard semi-permeable cellophane membrane. The membrane will be soaked in the release medium (simulated vaginal fluid 'SVF') overnight prior to its use. One gram solution of formulations will be weighed over the membrane in the dialytic tube. The prepared tube will be suspended in 100 ml freshly prepared SVF (simulated vaginal fluid ). The system will be placed into a constant temperature shaker water bath previously adjusted to 37 + 0.2 ºC and 50 rpm. Aliquots (1 ml) will be withdrawn from the release medium at each sampling time for up to 2 hours and the amount of the drug released will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* The selected patients had - vaginal candidiasis ,diagnosed by history of pruritus in addition to the characteristic discharge of vaginal candidiasis by vaginal examination

Exclusion Criteria:

* Women on other line of treatment as antimicrobial treatment either topical or systemic drugs within one month prior to the first clinical examination
* Known hypersensitivity for ketoconazole

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
measure effect of ketoconazole gel in treatment of vaginal candidiasis | ketoconazole used once daily for 3 days
  efficacy of ketoconazole gel by taking a vaginal swab for microbiological examination before treatment and another swab one week after treatment
improvement of patient complaint | one week
  improvement of vaginal symptoms and discharge

SECONDARY OUTCOMES:
rate of relapse | 2 weeks
  recurrence of symptoms and discharge (patient complaint )

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garcia Figueroa RG, Sauceda L, Ramirez Palacios D, Cruz Talonia F, Romero Cabello R. [Effectiveness and safety of ciclopirox olamine 1% vaginal cream versus terconazole 0.8% vaginal cream in the treatment of genital candidiasis]. Ginecol Obstet Mex. 2000 Apr;68:154-9. Spanish. PMID 10824446